CLINICAL TRIAL: NCT03135119
Title: Integrating Animal-Assisted Therapy Into Trauma-Focused Cognitive-Behavioral Therapy for Maltreated Youth: A Randomized Feasibility Trial
Brief Title: Integrating Animal-Assisted Therapy Into Trauma-Focused Cognitive-Behavioral Therapy for Maltreated Youth
Acronym: TF-CBT+AAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brian Allen, Associate Professor, Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006612; R21HD091887 (NIH)
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Child Abuse; Posttraumatic Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All individuals collecting and/or handling data will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TF-CBT (Active Comparator): Youth will receive standard Trauma-Focused Cognitive-Behavioral Therapy
  Interventions: Behavioral: TF-CBT
- TF-CBT+AAT (Experimental): Youth will received Trauma-Focused Cognitive-Behavioral Therapy with Animal-Assisted Therapy as an adjunct.
  Interventions: Behavioral: TF-CBT+AAT

INTERVENTIONS:
Behavioral: TF-CBT — TF-CBT is typically described as including 3 phases, each focusing on a common goal and encompassing a third of treatment (4 sessions). The first phase focuses on skills-building and includes psychoeducation, parenting skills training, relaxation skills training, affect modulation skills training, and cognitive coping skills training. The second phase involves focused gradual exposure activities, including construction of a narrative account of the child's maltreatment experiences and cognitive processing of maladaptive thoughts. The third phase emphasizes the child's mastery over environmental reminders of the maltreatment and includes sharing the trauma narrative with the caregiver, in vivo exposure to physical stimuli, and enhancing future development.
  Arms: TF-CBT
Behavioral: TF-CBT+AAT — TF-CBT, as described in the other arm, with animal-assisted therapy as an adjunct intervention. During the administration of TF-CBT, a certified service dog will be in the room and the participant may elect to interact with the dog as various points throughout the sessions.
  Arms: TF-CBT+AAT

SUMMARY:
This study will examine the incremental benefit of animal-assisted therapy (AAT) as an adjunct intervention when combined with Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT) for the treatment of maltreated youth. In addition, the development of therapeutic rapport and the intensity of stress experienced during treatment sessions will be examined as mediational mechanisms of treatment outcome. This project will help determine whether a larger study to test the beneficial effects of AAT for maltreated youth is feasible and warranted.

DETAILED DESCRIPTION:
The eventual goal of this line of research is to determine whether, and through what mechanisms, Animal-Assisted Therapy (AAT) is beneficial for the treatment of maltreated youth. The current project is a feasibility study to determine if larger clinical trials are warranted. The specific aims of the current study are (1) to examine whether the integration of AAT into standard Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT) enhances treatment effectiveness, (2) to evaluate the tolerability and feasibility of AAT when integrated into TF-CBT, and (3) to evaluate hypothesized mediational processes that may explain observed positive effects for the integration of AAT. Maltreated youth may display myriad emotional and behavioral symptoms; prominent among these is posttraumatic stress (PTS). TF-CBT is a well-established evidence-based treatment for PTS and other symptoms subsequent to child maltreatment and, therefore, is a suitable intervention for this trial. Sixty (60) maltreated youth (ages 6-17) displaying elevated PTS will be assigned to receive TF-CBT or TF-CBT+AAT using a blocked randomization procedure. The TF-CBT protocol is the standard twelve 90-minute sessions typically used in research trials. Youth in the TF-CBT+AAT condition will receive the standard protocol with a certified service dog present in the room for each session and the youth will be allowed to interact with the dog during session. A pre-post design will be used to ascertain whether the addition of AAT prompts greater PTS reduction as well as greater improvements in other outcomes, including internalizing symptoms, externalizing symptoms, and emotion regulation. Outcome metrics include caregiver and youth-reported objective measures, and respiratory sinus arrhythmia (RSA) assessed via an electrocardiogram (ECG) during both a resting and stress reactivity paradigm. Feasibility metrics assessed include treatment satisfaction, ability to implement the TF-CBT techniques with a dog in the room, treatment disrupting events attributable to the dogs, and whether the dogs experience significant stress as a result of their participation. Stress experienced by the dog will be determined through RSA, salivary cortisol, and behavioral responses. Two prominent hypotheses regarding the mechanism of effect for AAT will be examined. First, therapeutic rapport will be assessed at multiple increments to determine whether the presence of the dog improved the quality or efficiency of development of rapport. Second, RSA will be recorded for the youth during treatment sessions to determine if the presence of the dog yielded a lower intensity of stress during the sessions. Both therapeutic rapport and level of in-session stress will be examined as mediating variables to determine whether either explained enhanced treatment outcomes. To improve the methodological rigor of the study, data will be collected by research assistants blinded to the youth's treatment condition and the same clinicians will implement both treatment conditions, thereby eliminating clinician-specific effects on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A caregiver willing to participate with the youth
* An allegation of child maltreatment investigated by child protective services (CPS) or the police
* A raw score of ≥ 39 (borderline or clinical elevation) on the caregiver- report version of the UCLA PTSD Reaction Index for the DSM-5.

Exclusion Criteria:

* Severe developmental delays and/or psychiatric problems that necessitate a higher level of care for the child. An allegation of child maltreatment investigated by child protective services (CPS) or the police
* Intellectual deficits for the child (IQ < 80 on a cognitive screener)
* Caregiver inability to complete assessment measures due to psychiatric, cognitive, or other limitation
* The available caregiver is suspected or known to have perpetrated maltreatment
* A fear of dogs, a dog allergy, or any prior history of aggression toward animals for the child and/or caregiver

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Allen, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Medical Center-TLC Research and Treatment Center, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be stripped of individual identifiers prior to release for sharing. Data subsets will only be made available to other users under data-sharing agreements that provide for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Those wishing to access the data will need to directly contact the PI to complete the data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available starting in July, 2020, and will remain available for 5 years.
Access Criteria: Access to data will require:
  1. a commitment to using the data only for research purposes and not to identify any individual participant;
  2. a commitment to securing the data using appropriate computer technology;
  3. a commitment to destroying or returning the data after analyses are completed;
  4. A letter of approval from an applicable Institutional Review Board; and,
  5. A signed data usage agreement.

REFERENCES:
- [Derived] Shenk CE, Allen B, Dreschel NA, Wang M, Felt JM, Brown MP, Bucher AM, Chen MJ, Olson AE. Respiratory Sinus Arrhythmia Change during Trauma-Focused Cognitive-Behavioral Therapy: Results from a Randomized Controlled Feasibility Trial. Res Child Adolesc Psychopathol. 2022 Nov;50(11):1487-1499. doi: 10.1007/s10802-022-00946-w. Epub 2022 Jun 11. PMID 35689729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Youth were recruited to participate in this study, although caregivers are necessary to complete the treatment protocol and caregiver-report was a primary method of evaluating outcome. No measures were collected on caregiver functioning or outcomes. Recruitment numbers and outcomes are strictly related to the youth participants.
Period: Overall Study
Arm/Group | TF-CBT | TF-CBT+AAT
Started | 16 | 17
Completed | 11 | 14
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — COVID-19 Shutdown | 2 | 2

BASELINE CHARACTERISTICS:
Population: Caregivers completed measures reporting on the clinical outcomes of children and youth, but no baseline or outcome data were evaluated specific to caregiver functioning. All baseline and outcome data are child/youth-specific.
Groups:
- Total: Total of all reporting groups
Arm/Group | TF-CBT | TF-CBT+AAT | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.56 (3.35) | 12.0 (2.89) | 11.79 (3.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 9 | 12 | 21
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Scores on the UCLA Posttraumatic Stress Disorder Reaction Index
Description: This is a caregiver version of the measure designed to assess child/youth posttraumatic stress disorder (PTSD) symptoms. This is a 27-item questionnaire were the frequency of each item is reported using a scale ranging from 0 (Never) to 4 (Most Days), yielding a potential full scale score ranging from 0 to 108. For inclusion in this study, a score of at least 32 on the pre-treatment administration was required as this score denotes the "borderline" range for the measure. Lower scores indicate fewer PTSD symptoms are present.
Time Frame: Data were obtained at pre-treatment and every four weeks thereafter until the protocol was completed, **up to 13 weeks**. The last assessment completed, excluding the pre-treatment assessment, was considered post-treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TF-CBT | TF-CBT+AAT
Number analyzed (Participants) | 16 | 17
units on a scale
  Pre-treatment | 44.63 (12.38) | 39.5 (18.44)
  Post-treatment | 22.64 (16.43) | 35.85 (14.81)

2. Secondary Outcome: Change in Scores on the Strengths and Difficulties Questionnaire Emotional Symptoms Subscale
Description: The Strengths and Difficulties Questionnaire (SDQ) is a measure assessing the caregiver's observation of assorted emotional and behavioral concerns. This study utilized the "Emotional Symptoms" subscale, which collectively assesses symptoms of depression and anxiety. The subscale includes 5 items, each scored on a scale ranging from 0 (Never) to 2 (Certainly True). This results in possible total scores ranging from 0 to 10 with higher scores indicating a greater level of concern.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TF-CBT | TF-CBT+AAT
Number analyzed (Participants) | 16 | 17
units on a scale
  Pre-treatment | 6.5 (2.58) | 7.65 (2.0)
  Post-treatment | 4.0 (3.0) | 5.08 (1.85)

3. Secondary Outcome: Change in Scores on the Screen for Child Anxiety Related Disorders
Description: The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item measure where the youth self-reports on concerns related to various forms of anxiety. Answer options range from 0 (Not True or Hardly Ever True) to 2 (Very Often or Very True), resulting in a possible total score between 0 and 82 with higher scores indicating greater concerns.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TF-CBT | TF-CBT+AAT
Number analyzed (Participants) | 16 | 17
units on a scale
  Pre-treatment | 39.64 (18.04) | 35.47 (14.45)
  Post-treatment | 25.45 (19.17) | 31.62 (14.94)

4. Secondary Outcome: Change in Scores on the Moods and Feelings Questionnaire
Description: The Moods and Feelings Questionnaire (MFQ) is a 13-item measure that asks youth to report their own concerns with depression-related symptoms. Each item is answered with a 0 (Not True), 1 (Sometimes Ture), or 2 (True). The items are summed to create a total score that may range from 0 to 26, with higher scores denoting a greater level of depressive symptoms. .
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TF-CBT | TF-CBT+AAT
Number analyzed (Participants) | 16 | 17
units on a scale
  Pre-treatment | 9.13 (5.6) | 8.88 (4.69)
  Post-treatment | 5.91 (5.54) | 8.85 (6.12)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the course of the participant's participation in the study, which ran from the first assessment (i.e., pre-treatment) to their final attendance at a study related function (e.g., last treatment session attended, post-treatment assessment; **up to 13 weeks**)
Arm/Group | TF-CBT | TF-CBT+AAT
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03135119/Prot_SAP_000.pdf